CLINICAL TRIAL: NCT00005583
Title: A Randomized Trial of Adjuvant Treatment With Radiation Plus Chemotherapy Versus Radiation Alone in High Risk Endometrial Carcinoma
Brief Title: Radiation Therapy With or Without Chemotherapy in Treating Patients With High-Risk Endometrial Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nordic Society of Gynaecological Oncology - Clinical Trials Unit (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NSGO-EC9501; CDR0000067646 (Registry Identifier: PDQ (Physician Data Query)); EORTC-55991
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2006-11

CONDITIONS: Endometrial Cancer
Keywords: stage I endometrial carcinoma; stage II endometrial carcinoma; endometrial adenocarcinoma; endometrial papillary serous carcinoma; endometrial clear cell carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Cisplatin; Doxorubicin; Epirubicin; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether radiation therapy with chemotherapy is more effective than radiation therapy alone in treating high-risk endometrial cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy and chemotherapy to see how well they work compared to radiation therapy alone in treating patients with high-risk endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare relapse-free survival of patients with high-risk endometrial carcinoma treated in the adjuvant setting with either radiotherapy alone or radiotherapy and chemotherapy given sequentially.
* Compare overall survival of this patient population treated with these 2 adjuvant regimens.
* Evaluate the addition of chemotherapy to standard adjuvant radiotherapy, in terms of toxicity, in these patients.
* Study whether the pattern of relapse in these patients is influenced by the addition of chemotherapy to adjuvant radiotherapy.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to center and histologic type (serous papillary and clear cell vs all other types). Patients are randomized to 1 of 2 treatment arms.

All patients undergo hysterectomy with bilateral salpingooophorectomy and extirpation of macroscopic suspicious lymph nodes.

* Arm I: Within 7 weeks after surgery, patients begin radiotherapy.
* Arm II: Patients receive radiotherapy followed by or preceded by chemotherapy*. Patients receive cisplatin IV over 60 minutes and doxorubicin or epirubicin IV over 10-20 minutes on day 1. Treament repeats every 21 days for 4 courses.

NOTE: *If radiotherapy is preceded by chemotherapy, radiotherapy begins within 4 weeks after chemotherapy.

Patients are followed at 3 and 6 months and then every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 400 patients (200 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrial cancer of 1 of the following types:

  * Clear cell carcinoma
  * Serous papillary carcinoma
  * Undifferentiated (anaplastic) carcinoma
  * Poorly differentiated (FIGO grade 3) adenocarcinoma with infiltration to more than half the myometrial thickness
* No small cell carcinoma with neuroendocrine differentiation
* Primary in FIGO surgical stage I or occult stage II
* No spread of disease outside the uterine corpus except to pelvic lymph nodes

  * No spread of disease to para-aortic lymph nodes
* Positive peritoneal washings allowed
* No preoperative macroscopic tumor involvement of the cervix

  * Microscopic tumor involvement of the cervix on histopathological evaluation of the operative uterine specimen allowed

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Adequate bone marrow function
* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Adequate hepatic function

Renal:

* Adequate renal function
* Creatinine no greater than 1.4 mg/dL

Pulmonary:

* Adequate pulmonary function

Other:

* Not pregnant or nursing
* Fit to receive combination chemotherapy
* No other malignancy except basal cell or squamous cell skin cancer
* No uncontrolled or potentially active site of infection (e.g., fistula or abscesses)
* No other concurrent condition that would produce a substantial increase in risk for complications from radiotherapy
* No other concurrent condition that would interfere with adequate follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior preoperative irradiation

Surgery:

* No prior extensive abdominal surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2000-01; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival
Relapse-free survival

SECONDARY OUTCOMES:
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar B. Kristensen, MD, PhD, Study Chair — Norwegian Radium Hospital; Carlos F. de Oliveira, MD, PhD — Hospitais da Universidade de Coimbra (HUC)
Locations (23):
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - U.Z. Gasthuisberg, Leuven
- Centre Henri Becquerel, Rouen, France
- Ireland (2):
  - Coombe Women's Hospital, Dublin
  - St. James's Hospital, Dublin
- Italy (4):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Azienda Ospedaliera Di Parma, Parma
  - Fondazione I.R.C.C.S. Policlinico San Matteo, Pavia
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
- Norwegian Radium Hospital, Oslo, Norway
- Medical University of Gdansk, Gdansk, Poland
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Groote Schuur Hospital, Cape Town, South Africa
- Spain (2):
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
- United Kingdom (3):
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Centre for Cancer Research and Cell Biology at Belfast City Hospital, Belfast, Northern Ireland
  - Western Infirmary, Glasgow, Scotland

REFERENCES:
- [Background] Hogberg T, Signorelli M, de Oliveira CF, Fossati R, Lissoni AA, Sorbe B, Andersson H, Grenman S, Lundgren C, Rosenberg P, Boman K, Tholander B, Scambia G, Reed N, Cormio G, Tognon G, Clarke J, Sawicki T, Zola P, Kristensen G. Sequential adjuvant chemotherapy and radiotherapy in endometrial cancer--results from two randomised studies. Eur J Cancer. 2010 Sep;46(13):2422-31. doi: 10.1016/j.ejca.2010.06.002. Epub 2010 Jul 7. PMID 20619634
- [Result] Hogberg T, Rosenberg P, Kristensen G, et al.: A randomized phase-III study on adjuvant treatment with radiation (RT) ± chemotherapy (CT) in early-stage high-risk endometrial cancer (NSGO-EC-9501/EORTC 55991). [Abstract] J Clin Oncol 25 (Suppl 18): A-5503, 274s, 2007.